CLINICAL TRIAL: NCT01604694
Title: Ultrasound-guided Transversus Abdominis Plane Block for Analgesia After Abdominoplasty: Randomized- Controlled- Trial Double Blind Monocentric Study, Against Placebo
Brief Title: Ultrasound-guided Transversus Abdominis Plane Block for Analgesia After Abdominoplasty
Acronym: TAPlastie
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2011/10
Record Dates: First submitted 2012-05-15; First posted 2012-05-24 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Abdominoplasty; Transversus Abdominis Plane (TAP) Block
Keywords: Abdominoplasty; Transversus Abdominis Plane (TAP) Block; levobupivacaine; Placebo
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP Block with levobupivacaïne (Experimental)
  Interventions: Procedure: TAP Block
- TAP Block with Placebo (Placebo Comparator)
  Interventions: Procedure: TAP Block

INTERVENTIONS:
Procedure: TAP Block — An Ultra Sound-guided TAP block is performed after induction of general anesthesia prior to surgical incision. The syringes containing either saline 20 ml (placebo group) or levobupivacaine 20 ml are prepared by the hospital pharmacy under aseptic conditions.

SUMMARY:
Abdominoplasty is a major cosmetic surgery with a painful post operative period. Recently more and more anaesthetists are turning to regional analgesia for anterior abdominal wall surgery namely the Transversus Abdominis Plane (TAP) Block with or without ultrasound guidance.

The aim of this study is to evaluate the analgesic effect of TAP block ultrasound guided in post operative period of abdominoplasty.

DETAILED DESCRIPTION:
To determine if TAP block have an analgesic effect in post operative period of abdominoplasty this study was made versus placebo: one group of patients will have a TAP block of levobupivacaine, the second group will have a TAP block with placebo before the surgery. Patient follow up includes data collected before surgery (at pré anesthesic visit and just before surgery) and data collected immediately after surgery (at post operative time) and at distance of the surgery (15 days and 3 months after the surgery). The principal aim is to show if TAP block have an analgesic effect in post operative period after abdominoplasty. To answer this question we will compare opioid intake during the two days after the surgery between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA1 or 2 patients
* Undergoing abdominoplasty surgery in Centre François Xavier Michelet at Bordeaux University hospital
* Age >18 years old
* Patient agreement by signing an informed consent

Exclusion Criteria:

* Psychiatric or neurological disease
* Contraindication to regional anesthesia (haemostatic disorders, infection near to insertion point)
* Double surgery
* Long term opioid therapy
* Pregnancy or breast-feeding
* Allergy to any drug used in anesthesic or surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Opioid consumption during 24 hours after the surgery | 24 hours after surgery

SECONDARY OUTCOMES:
Quality of analgesia | Until 48 hours after surgery
  Evaluated by opioid consumption, visual scale assessment of pain by patient, occurrence of specific adverse events (nausea, vomiting, somnolence, pruritus...)
Early rehabilitation : hour of first rising, six-minute walk test at 3days and at discharge | Until discharge, up to 8 days after surgery
Evaluation of Neuropathic pain, pain thresholds, hyperalgesia area | 15 days and 3 month after surgery
Health - related quality of life preoperative and at 3 months post operatively | Just before and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD, Study Chair — USMR, University Hospital Bordeaux
Locations (1):
- CHU de Bordeaux, Centre François-Xavier Michelet, Bordeaux, France